CLINICAL TRIAL: NCT06893783
Title: A Phase II Trial of Tarlatamab, a DLL3-targeted Bispecific T-cell Engager, in Patients With Advanced Extrapulmonary Neuroendocrine Carcinoma (DeLLight)
Brief Title: Efficacy and Safety Evaluation of Tarlatamab in Advanced Extrapulmonary Neuroendocrine Carcinoma Patients
Acronym: DeLLight
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inkeun Park (Other)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, Inkeun Park, Clinical Associate professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeLLight
Record Dates: First submitted 2025-02-21; First posted 2025-03-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Carcinomas (NEC); Neuroendocrine Carcinoma of Pancreas; Neuroendocrine Carcinoma of Prostate
Keywords: extrapulmonary neuroendocrine carcinoma; Tarlatamab; bispecific t-cell engager; DLL3
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — DLL3 protein, human

STUDY DESIGN:
Intervention Model Description: The study will be divided into a gastrointestinal and pancreatic-biliary cohort and a genitourinary cohort; however, the dosage, frequency, duration, and administration route of the investigational drug will remain the same as outlined below.
  Tarlatamab
  1 mg step dose on cycle 1 day 1 10 mg target dose starting cycle 1 day 8, cycle 1 day 15, and every 2weeks thereafter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All patient (Experimental): The study will be divided into a gastrointestinal and pancreatic-biliary cohort and a genitourinary cohort; however, the dosage, frequency, duration, and administration route of the investigational drug will remain the same as outlined below.
  Tarlatamab
  1 mg step dose on cycle 1 day 1 10 mg target dose starting cycle 1 day 8, cycle 1 day 15, and every 2weeks thereafter
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — 1 mg step dose on cycle 1 day 1 10 mg target dose starting cycle 1 day 8, cycle 1 day 15, and every 2weeks thereafter
  Other Names: Delta-like ligand 3 (DLL3) Bispecific T-Cell Engager

SUMMARY:
This is a phase 2 single-arm, open-label clinical trial designed to evaluate the efficacy and safety of tarlatamab in patients with relapsed extrapulmonary neuroendocrine carcinoma (EPNEC) who have previously received platinum-based first-line chemotherapy. Participants will receive tarlatamab on Cycle 1 Day 1 (C1D1), Day 8 (C1D8), and Day 15 (C1D15), followed by administration every two weeks thereafter. No placebo control is included in this study.

DETAILED DESCRIPTION:
1. study rationale Extrapulmonary neuroendocrine carcinomas (EPNECs) are rare, aggressive malignancies with poor prognosis, lacking established second-line treatments. First-line therapy, adapted from small cell lung cancer (SCLC), consists of platinum-based chemotherapy, but responses are short-lived, and salvage options offer limited benefit (response rates 10-30%, overall survival 5-7 months).

   Delta-like ligand 3 (DLL3) is highly expressed in EPNECs, making it a promising therapeutic target. Tarlatamab, a DLL3-targeting bispecific T cell engager (BiTE), has demonstrated durable antitumor activity in relapsed SCLC. Given its efficacy in DLL3-expressing tumors, tarlatamab may provide a novel treatment option for EPNECs.
2. Study Design This is an open-label, single-arm, multi-center, phase 2 study that will evaluate efficacy and safety of tarlatamab (AMG 757) for the treatment of subjects with extrapulmonary neuroendocrine carcinomas (EPNECs) who have progressed after 1 prior line of platinum-containing therapy. The study will be composed of 2 cohorts; cohort 1 (gastrointestinal and pancreaticobiliary NEC) and cohort 2 (genitourinary NEC).

   The study consists of a 21-day screening period, a treatment period, a safety follow-up (SFU) visit, and a long-term follow-up (LTFU) period.
3. The primary objective of the study is to assess the efficacy of tarlatamab based on the objective response rate (ORR) as determined by investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. The primary estimand focuses on the proportion of participants achieving a partial or complete response.

   A secondary objective is to evaluate progression-free survival (PFS), defined as the time from treatment initiation until disease progression or death.
4. Intervention Details

Participants will receive tarlatamab via intravenous (IV) infusion according to the following schedule:

Cycle 1:

Day 1 (C1D1): 1 mg IV over 60 minutes Day 8 (C1D8): 10 mg IV over 60 minutes Day 15 (C1D15): 10 mg IV over 60 minutes Subsequent Cycles: 10 mg IV every two weeks There is no placebo in this study.

ELIGIBILITY:
Inclusion Criteria:

- Subject has provided informed consent prior to initiation of any study specific activities/procedures.

* Age ≥19 years at the time of signing the informed consent.
* Histologically confirmed relapsed/refractory extra-pulmonary neuroendocrine carcinoma. Neuroendocrine carcinoma includes small cell carcinoma, large cell carcinoma, and mixed histology of neuroendocrine and other histology (e.g., adenoneuroendocrine carcinoma, urothelial carcinoma with neuroendocrine component). In patients with prostate cancer, treatment-emergent neuroendocrine carcinoma (initially adenocarcinoma, but transdifferentiate into neuroendocrine carcinoma after androgen deprivation therapy) will be permitted.
* Cohort 1 (gastrointestinal and pancreaticobiliary cohort): cancers originated from stomach, small intestine, colorectal, pancreas, or bile ducts.
* Cohort 2 (genitourinary cohort): cancers originated from prostate, bladder, ureter, urethra, or kidney.
* Subject has progressed or recurred following 1 platinum-based regimen:
* documented first disease progression must be during or following first-line platinum-based systemic chemotherapy. For patients with prostate cancer, especially in cases with treatment-emergent neuroendocrine carcinoma, platinum-based chemotherapy will not need to be the first line therapy.

  * patients who received treatment for localized disease who recur are eligible
  * patients who received adjuvant Platinum-Etoposide (EP) after resection of their primary tumor who recur are eligible
* Measurable disease as defined per RECIST 1.1 within the 21-day screening period.

  • Screening scans performed as SOC(Standard of Care) and prior to informed consent, may be used to confirm subject eligibility if completed within the 21-day screening period, provided that informed consent for the use of these scans is obtained prior to any transfer of data.
  * In patients with prostate cancer, patients without RECIST-defined measurable lesion can be included, if disease can be evaluated with Prostate Cancer Working Group(PCWG)-3 criteria.
* Eastern Cooperative Oncology Group (ECOG) PS(Performance Status) of 0 - 2.
* Minimum life expectancy of 12 weeks.
* Adequate organ function, defined as follows:

  • Hematological function: Absolute neutrophil count ≥ 1.5 x 10^9 /L Platelet count ≥ 100 x 10^9/L Hemoglobin > 9 g/dL (90 g/L)

  • Coagulation function: Prothrombin Time (PT)/International Normalized Ratio (INR) and Partial Thromboplastin Time (PTT) or activated Partial Thromboplastin Time (APTT) ≤ 1.5 x institutional upper limit of normal (ULN) except for subjects undergoing new class anticoagulant therapy (eg, Edoxaban), stable dose for 2 weeks required prior to enrollment.

  • Renal function: estimated glomerular filtration rate (eGFR) based on Modification of Diet in Renal Disease (MDRD) calculation ≥ 30 mL/min/1.73 m^2 or creatinine clearance ≥ 30 mL/min as determined by Cockcroft-Gault equation (Cockcroft and Gault 1976)

  • Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN (or <5 x ULN for subjects with liver involvement) total bilirubin (TBL) <1.5 x ULN (<2 x ULN for subjects with liver involvement) (except participants with Gilbert syndrome who must have total bilirubin <3.0 mg/dL)

  • Pulmonary function: no clinically significant pleural effusion. Pleural effusion managed with indwelling pleural catheter (eg, PleurX) are allowed baseline oxygen saturation >90% on room air

  • Cardiac function: cardiac ejection fraction ≥50%, no clinically significant pericardial effusion as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan, and no clinically significant electrocardiogram (ECG) findings Provision of evaluable tumor samples for central testing (archival or in-study biopsy)

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases:

  • Subjects with treated brain metastases are eligible provided the following criteria are met:
* Subject is asymptomatic from brain metastases
* Whole brain radiation or surgery was completed at least 2 weeks prior to first dose of study treatment (stereotactic radiosurgery completed at least 7 days prior to first dose of study treatment)
* Any CNS disease is clinically stable, subject is off steroids for CNS disease for at least 5 days (unless steroids are indicated for a reason unrelated to CNS disease), and subject is off or on stable doses of anti-epileptic drugs at least 14 days prior to first dose of study treatment • Subjects with untreated brain metastases that are asymptomatic and do not require corticosteroids, nor local therapy per investigators standard of practice are allowed Diagnosis or evidence of leptomeningeal disease.

Prior history of immune checkpoint inhibitors resulting in:

* Any severe or life-threatening immune-mediated adverse event, History of immune-mediated encephalitis or other immune-mediated CNS event (any grade)
* Grade ≥ 2 immune-mediated recurrent pneumonitis, Infusion-related reactions leading to permanent discontinuation of immunotherapy agent Exception: Subjects with a history of immune checkpoint inhibitor-induced endocrinopathy which is clinically stable on replacement therapy.

  * Active autoimmune disease that has required systemic treatment (except replacement therapy) within the past 2 years or any other diseases requiring immunosuppressive therapy while on study.
  * History of solid organ transplantation.
  * History of other malignancy within the past 2 years, with the following exceptions:
* low-risk malignancy treated with curative intent and with no known active disease present for ≥ 1 year before enrollment and believed to be at low risk for recurrence per investigator discretion.
* adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, cervical carcinoma in situ without evidence of disease, breast ductal carcinoma in situ without evidence of disease.
* prostatic intraepithelial neoplasia without evidence of prostate cancer. (For non-prostate cancer patient)
* adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.

  * Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association > class II) within 12 months prior to first dose of study treatment (Section 11.9).
  * History of arterial thrombosis (eg, stroke or transient ischemic attack) within 12 months prior to first dose of study treatment.
  * Presence/history of viral infection: Human immunodeficiency virus (HIV) infection
* Subjects with HIV infection on antiviral therapy and undetectable viral load are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on study per local or institutional guidelines, Active hepatitis C infection (subjects with detectable hepatitis C antibody [HCV Ab] and HCV RNA viral load above the limit of quantification),
* Subjects with presence of HCV Ab and HCV RNA viral load below the limit of quantification (HCV RNA negative) with or without prior treatment are allowed Active hepatitis B infection (presence of hepatitis B surface antigen [HBsAg] and hepatitis B virus [HBV] DNA viral load above the limit of quantification [HBV DNA positive])
* Subjects with resolved HBV infection defined as absence of HBsAg and presence of HBV core antibody (anti-HBc) followed by an HBV DNA viral load below the limit of quantification (HBV DNA negative) are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.
* Subjects with chronic HBV infection inactive carrier state defined as presence of HBsAg and HBV DNA viral load below the limit of quantification [HBV DNA negative] are allowed, with a requirement for regular monitoring for reactivation for the duration of treatment on the study and assessing the need for HBV prophylaxis therapy per local or institutional guidelines.

Receiving systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days prior to first dose of study treatment:

* Prophylactic dexamethasone required by the protocol and any anti-emetic therapies are allowed
* Low-dose corticosteroids (prednisone ≤10 mg per day or equivalent is permitted during the trial)

  * Subject with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.
  * Evidence of interstitial lung disease or active, non-infectious pneumonitis.
  * Prior therapy with tarlatamab
  * Prior therapy with any selective inhibitor of the DLL3 pathway.
  * Subject received more than 2 prior systemic therapy regimens for EPNECs. In patients with treatment-emergent prostate neuroendocrine carcinoma, treatments given before histological confirmation of neuroendocrine cancer (e.g., androgen deprivation therapy, androgen receptor targeted agents such as enzalutamide and abiraterone, and docetaxel) are not considered as previous treatment for metastatic/recurrent EPNEC.
  * Prior anti-cancer therapy within 21 days prior to first dose of study treatment. Exceptions:
* Subjects who received conventional chemotherapy are eligible if at least 14 days have elapsed and if all treatment-related toxicity has been resolved to grade ≤ 1, or to levels dictated in the eligibility criteria, before first dose of study treatment, with the exception of alopecia or toxicities considered irreversible (defined as having been present and stable for >30 days) which are not otherwise described in the exclusion criteria.
* Prior palliative radiotherapy must have been completed at least 7 days before the first dose of study treatment.

  * Receiving anti-cancer therapy such as chemotherapy, immunotherapy, or targeted therapy. Patients who are receiving adjuvant hormonal therapy for resected breast cancer may be eligible (refer also to exclusion related to history of other malignancies). Additionally, in patients with treatment-emergent prostate neuroendocrine carcinoma, continuation of androgen deprivation therapy is permitted.
  * Any herbal or prescription/non-prescription medications known to inhibit membrane transporters P-glycoprotein (P-gp) and/or breast cancer resistance protein (BCRP) within 7 days prior to the first dose of study treatment.

Any herbal or prescription/non-prescription medications known to be moderate or strong inhibitors of cytochrome P450 3A (CYP3A) enzymes (including but not limited to clarithromycin, itraconazole, ketoconazole) within 7 days prior to the first dose of study treatment.

* Any herbal or prescription/non-prescription medications known to be moderate or strong inducers of CYP3A enzymes within 28 days prior to first dose of study treatment.
* Subjects who have reached the limit dose of prior treatment with cardiotoxic drugs such as other anthracyclines.
* Major surgical procedures within 28 days prior to first dose of study treatment.

Treatment with live virus, including live-attenuated vaccination, within 14 days prior to the first dose of study treatment. Inactive vaccines (eg, non-live or non-replicating agent) and live viral non-replicating vaccines (eg, Jynneos for Monkeypox infection) within 3 days prior to first dose of study treatment.

* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Female subjects of childbearing potential unwilling to use protocol specified method of contraception see Appendix 5 (Section 11.5) during treatment and for an additional 60 days after the last dose of tarlatamab.
* Female subjects who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of tarlatamab
* Female subjects planning to become pregnant or donate eggs while on study through 60 days after the last dose of tarlatamab
* Female subjects of childbearing potential with a positive pregnancy test assessed at screening by a serum or urine pregnancy test.
* Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 60 days after the last dose of tarlatamab.
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of tarlatamab
* Male subjects unwilling to abstain from donating sperm during treatment and for an additional 60 days after the last dose of tarlatamab Subject has known sensitivity or is contraindicated to any of the products or components to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures
* History or evidence of any other clinically significant disorder, condition or disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From the date of first dose until the date of the first confirmed objective response (PR or CR) per RECIST v1.1, assessed up to 36 months
  defined as the percentage of participants who have a partial response or complete response based on investigator assessment per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  defined as time from treatment initiation until disease progression or death from any cause, whichever occurs first for all subjects. Progression will be based on investigator assessment of disease response per RECIST 1.1
Overall Survival(OS) | From the date of the safety follow-up visit for up to 36 months after the last subject is enrolled or 1 year after the last subject's final dose of study treatment, whichever is later
  defined as time from treatment initiation until death from any cause
Duration of response (DOR) | From the date of the first recorded objective response (partial response [PR] or complete response [CR]) for up to 36 months, until the first documented date of disease progression or death from any cause, whichever occurs first.
  defined as the time from the first documentation of OR until the first documentation of disease progression or death due to any cause, whichever occurs first. Only subjects who have achieved OR will be evaluated for DOR

CONTACTS AND LOCATIONS:
Overall Officials: Inkeun Park, M.D, Ph D, Principal Investigator — Asan Medical Center
Locations (4):
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No